CLINICAL TRIAL: NCT06144476
Title: Study of Inflammatory and Physiological Profiles of Healthy and Diseased Lung
Acronym: RETAIN
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: 322540
Record Dates: First submitted 2023-08-22; First posted 2023-11-22 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: COPD; Asthma; Airway Disease
Keywords: Airway Disease; Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All samples will be collected for exploratory research including future genetic/DNA research.
  Sputum:
  Phosphate buffered saline (PBS) and dithiothreitol (DTT) sputum supernatant, Sputum cell cytospins, Sputum cellular pellet
  Nasal:
  Nasosorption swabs, Nasopharyngeal swabs, Nasal lavage, Nasal brushings
  Breath:
  Exhaled Breath
  Blood:
  Whole blood, Blood cells, Serum/plasma
  Bronchoscopy:
  Bronchial biopsies, Bronchial lavage, Bronchosorption swabs, Bronchial brushings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Airways Disease: Patients with or suspected airways disease including COPD or asthma
- Healthy Volunteers: Participants with no significant illness

SUMMARY:
There are over 700,000 UK hospital admissions every year with lung disease symptoms. Two of the most common lung diseases contributing to these numbers are asthma and chronic obstructive pulmonary disease (COPD). The immunopathology of these diseases is not fully understood. Matched samples from the respiratory tract and circulation will be used to identify immune patterns throughout the respiratory system to elucidate the immunopathology of airway disease.

DETAILED DESCRIPTION:
In this observational study, we will be enrolling patients with diagnosed or suspected airways disease who are over 18 years old, as well as age matched healthy volunteers with no significant illness. Participants will be asked if they consent to enter the study, invited at clinically relevant time points (treatment change, disease exacerbation etc.) and to optional bronchoscopy visits. It is expected that participants will be seen yearly with any additional exacerbation/treatment visits also recorded. Research visits will occur at King's College London and the Guys and St Thomas' NHS Foundation Trust (GSTFT), with all bronchoscopy visits occurring within GSTFT

1. Disease specific questionnaires.
2. Lung function tests including spirometry or oscillometry (if not performed previously within 6 months)
3. Sputum collection
4. Nasal sampling including nasosorption, nasal brushing, nasal lavage, or nasopharyngeal swabs
5. Exhaled breath
6. Blood samples (<6 tablespoons)

   Optional
7. Bronchoscopy involving a flexible fibreoptic camera passed into the lungs to collect bronchoalveolar lavage, bronchosorption, bronchial brushings and bronchial biopsies.
8. To repeat these procedures at later time - expected once per year or at times of clinically relevant changes

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Aged 18 years or above
* Patient: known or suspected airway disease
* Healthy volunteer: considered to be in good health with no significant comorbidity (immune disorder, cancer etc.)

Exclusion Criteria:

* Known or suspected current pulmonary tuberculosis, HIV (human immunodeficiency virus), Hepatitis B Virus, Hepatitis C Virus.
* Surgery within the preceding 6 weeks
* Participants who are pregnant
* History of psychiatric, medical, or surgical disorders that in the opinion of the chief investigator may interfere with sample collection, undergo a bronchoscopy, or may compromise study completion or data collection
* Alcohol or recreational drug abuse
* Diagnosis of immunodeficiency requiring treatment
* Unable to provide written informed consent
* Unable to read or write English
* Be considered, in the opinion of the investigator, to be an unsuitable candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include patients diagnosed or with suspected COPD and asthma. The study will include both current and former smokers.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Blood samples for presence of airway disease immune endotypes | 6 years
  Blood samples taken to assess inflammatory mediators to determine airway disease severity. Physiological and inflammatory characterisation of participants with known or suspected airway disease at stable state, compared to healthy volunteers with the aim to identify distinct immune endotypes in airways disease

SECONDARY OUTCOMES:
Blood samples for stability of airway disease immune endotypes | 6 years
  To assess the stability of blood inflammatory mediators to identify continuing airway disease endotypes. Longitudinal analysis of physiological and inflammatory characteristics in participants with known or suspected airway disease at stable state, compared to healthy volunteers over time.

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, Prof, Principal Investigator — GSTT and KCL
Locations (1):
- Guy's & St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No